CLINICAL TRIAL: NCT04865341
Title: Optimizing an IMB-guided Intervention to Support HIV Self-testing and PrEP Uptake Among YMSM: A Pilot Factorial RCT
Brief Title: IMB-guided Intervention to Encourage PrEP Uptake Among Young Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Steven A John, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PRO34897
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV testing; HIV pre-exposure prophylaxis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMB (Experimental): Individuals randomized to this arm will receive a behavioral intervention based on the Information-Motivation-Behavior (IMB) model designed to increase HIV self-testing, among other protective behaviors.
  Interventions: Behavioral: IMB
- Information-Only Control (Other): Attention-matched comparison condition (information-only)
  Interventions: Behavioral: Information-Only Control

INTERVENTIONS:
Behavioral: IMB — Intervention content will be focused on the Information-Motivation-Behavioral Skills (IMB) model. We plan to incorporate previously developed content as much as possible and will include professionally produced videos about HIV testing and PrEP and other resources. We believe our approach of guiding YMSM through intervention modules based on theory will help improve content retention/use and ultimately influence constructs posited to result in behavior change. We foresee using multiple forms of attention-matched material, media, and programming to engage (and retain engagement) of YMSM throughout the brief single-session intervention (45-60 minutes).
  Arms: IMB
Behavioral: Information-Only Control — Intervention content will be focused on the information construct of the Information-Motivation-Behavioral Skills (IMB) model. We plan to incorporate previously developed content as much as possible and will include professionally produced videos about HIV testing and PrEP and other resources. We believe our approach of guiding YMSM through intervention modules based on theory will help improve content retention/use and ultimately influence constructs posited to result in behavior change. We foresee using multiple forms of attention-matched material, media, and programming to engage (and retain engagement) of YMSM throughout the brief single-session intervention (45-60 minutes).
  Arms: Information-Only Control

SUMMARY:
The proposed study will involve adolescent (17-24 years old) men who have sex with men (described as YMSM hereafter) who meet eligibility criteria to participate in each study. Prospective study candidates will receive a copy of the IRB-approved informed consent forms and, if they choose to participate, will provide consent before enrollment into this study. Involvement of human subjects is detailed in the Research Strategy portion of this proposal, Recruitment and Retention Plan, and Protection of Human Subjects sections. Briefly, investigators will develop and pilot a randomized controlled trial (RCT) to support HIV self-testing (HIVST) and pre-exposure prophylaxis (PrEP) uptake. Intervention content will be focused on constructs of the Information-Motivation-Behavioral Skills (IMB) model. To reduce cost and increase feasibility, investigators plan to incorporate previously developed content as much as possible-investigators see integration of this content as a major strength. Investigators will include professionally produced videos about HIV testing and PrEP and other resources including the geo-targeted directories to find clinic settings that offer HIV testing and PrEP, all of which are publicly available. Investigators believe our approach of guiding YMSM through intervention modules based on theory will help improve content retention/use and ultimately influence constructs posited to result in behavior change. Investigators foresee using multiple forms of attention-matched material, media, and programming to engage (and retain engagement) of YMSM throughout the brief single-session intervention (45-60 minutes). Intervention content is subject to change depending on feedback from focus groups, survey results, YAB feedback, and usability testing. Primary endpoints of this study include HIVST and PrEP uptake, including stage of change towards HIVST and PrEP uptake. Secondary outcomes include changes in IMB model indicators (e.g., HIV prevention knowledge).

DETAILED DESCRIPTION:
The research activity designated as a clinical trial is our pilot RCT where investigators will then enroll 120 YMSM and randomly assign individuals to one of two experimental groups: (1) information-only (I), and (2) information + motivation + behavioral skills (IMB). Randomization will be blinded using Qualtrics, and randomization will occur in a ratio of 1:1 between the two groups. Individuals assigned to group 1 will receive attention-matched information-only filler content (e.g., information about physical activity and diet), but note that group (1) information-only will still receive HIVST and PrEP related information. Intervention content will be based upon the formative research. After completion of the baseline survey, randomization, and intervention, participants will be followed for a period of three months. Individuals will be surveyed at 1- and 3-months post intervention to assess our primary endpoints of HIVST and PrEP uptake. Preliminary impact will be assessed using within- and between-subjects analyses. First, investigators will test the performance of randomization by chi-squared comparisons and ANOVAs for categorical and continuous variables, respectively. Second, investigators will test for differential attrition by treatment group at 1- and 3-month follow-up assessments. Third, investigators will assess post-intervention HIV testing and PrEP uptake using factorial logistic regressions to determine between-group differences, adjusting for any breakdowns in randomization or differential attrition. Fourth, investigators will test for changes in stage of change indicators by randomized group, time, and group*time interaction, with similar adjustment procedures, using GEE; this analysis will help us determine a trend towards HIVST or PrEP uptake were investigators to extend the length of follow-up. Power: Our study has 80% power to detect a ½ stage average difference (d = 0.68; α = 0.05) on the PrEP cascade comparing the three experimental groups combined to the information-only control assuming 80% retention. As the purpose of this study is to pilot the RCT, investigators have not powered this study to determine differences between the experimental group compared to the control group (which is planned for the full RCT in a future R01). Finally, investigators will conduct within-subjects tests comparing baseline and follow-up IMB construct scale scores stratified by group as an evaluation of internal validity (i.e., did the interventions have an effect on the targeted constructs?).

ELIGIBILITY:
Inclusion Criteria:

1. 17-24 years old;
2. Individuals who self-identify as male (including transgender men) and report any male sexual partners in the past 6 months;
3. Resident of the US based on home address;
4. HIV-negative or unknown status based on self-report; and
5. Self-reported risk for HIV (based on CDC criteria for PrEP use) defined as reporting any of the following in the past six months:

   1. Bacterial STI
   2. Condomless anal sex (CAS) with a casual male sexual partner
   3. CAS with an HIV-positive or unknown status main partner
   4. CAS with an HIV-negative main partner who reports CAS with other male partners.

Exclusion Criteria:

1. Current PrEP use;
2. Unstable, serious psychiatric symptoms;
3. Currently suicidal/homicidal; and
4. Evidence of gross cognitive impairment.

Ages: 17 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the number of self-reported HIV self-tests | 3 months
  Self-reported self-administration of HIV testing within the past 3 months (i.e., since baseline assessment).
PrEP uptake | 3 months
  Self-reported PrEP uptake

CONTACTS AND LOCATIONS:
Overall Officials: Steven A John, MPH, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] John SA, Lopez-Rios J, Starks TJ, Rendina HJ, Grov C. Willingness to Distribute HIV Self-Testing Kits to Recent Sex Partners Among HIV-Negative Gay and Bisexual Men and an Examination of Free-Response Data from Young Men Participating in the Nationwide Cohort. Arch Sex Behav. 2020 Aug;49(6):2081-2089. doi: 10.1007/s10508-020-01752-5. Epub 2020 Jun 3. PMID 32495242
- [Background] John SA, Walsh JL, Quinn KG, Cho YI, Weinhardt LS. Testing the Interpersonal-Behavior model to explain intentions to use patient-delivered partner therapy. PLoS One. 2020 May 20;15(5):e0233348. doi: 10.1371/journal.pone.0233348. eCollection 2020. PMID 32433680
- [Background] John SA, Quinn KG, Pleuhs B, Walsh JL, Petroll AE. HIV Post-Exposure Prophylaxis (PEP) Awareness and Non-Occupational PEP (nPEP) Prescribing History Among U.S. Healthcare Providers. AIDS Behav. 2020 Nov;24(11):3124-3131. doi: 10.1007/s10461-020-02866-6. PMID 32300991
- [Background] Quinn KG, Zarwell M, John SA, Christenson E, Walsh JL. Perceptions of PrEP Use Within Primary Relationships Among Young Black Gay, Bisexual, and Other Men Who Have Sex with Men. Arch Sex Behav. 2020 Aug;49(6):2117-2128. doi: 10.1007/s10508-020-01683-1. Epub 2020 Apr 2. PMID 32240437
- [Background] Pleuhs B, Quinn KG, Walsh JL, Petroll AE, John SA. Health Care Provider Barriers to HIV Pre-Exposure Prophylaxis in the United States: A Systematic Review. AIDS Patient Care STDS. 2020 Mar;34(3):111-123. doi: 10.1089/apc.2019.0189. Epub 2020 Feb 28. PMID 32109141